CLINICAL TRIAL: NCT05376644
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Using 99mTc-ADAPT6 and 99mTc-DARPinG3 in HER2-positive Breast Cancer Patients Before System (Chemo/Targeted) Therapy.
Brief Title: Molecular Imaging of HER2 Expression in HER2-positive Breast Cancer Using 99mTc-ADAPT6 vs 99mTc-DARPinG3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99mTc-ADAPT6 vs 99mTc-DARPinG3
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Female
Keywords: 99mTc-ADAPT6; 99mTc-DARPinG3; Breast Cancer; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Diagnostic Test: ADAPT6-SPECT and DARPinG3-SPECT Diagnostic SPECT for HER2-positive Breast Cancer primary tumour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2 positive breast cancer patients (Experimental): Maximum (15) evaluable subjects with HER2-positive status in primary tumour before chemo/targeted therapy have to be enrolled in the study. Subjects withdrawn from the study for any reason will be replaced
  Interventions: Drug: 99mTc-ADAPT6; Drug: 99mTc-DARPinG3

INTERVENTIONS:
Drug: 99mTc-ADAPT6 — One single injection of 99mTc-ADAPT6, followed by gamma camera imaging 2 hours after injection.
  Other Names: SPECT
Drug: 99mTc-DARPinG3 — One single injection of 99mTc-DARPinG3, followed by gamma camera imaging 4 hours after injection.
  Other Names: SPECT

SUMMARY:
An open-label, single center study with 99mTc-ADAPT6 and 99mTc-DARPinG3 SPECT and biopsies of primary tumour in HER2-positive Breast Cancer before system (chemo/targeted) therapy, where the primary endpoint of the study is to compare imaging properties of 99mTc-ADAPT6 and 99mTc-DARPin G3 SPECT in HER2-positive breast cancer patients.

DETAILED DESCRIPTION:
The primary objectives are:

Compare SPECT/CT imaging properties of 99mTc-ADAPT6 and 99mTc-DARPin G3 in HER2-positive primary tumour of breast cancer patients before system (chemo/targeted) therapy.

The secondary objectives are:

To compare the SPECT/CT tumor imaging data with the data concerning HER2 expression obtained by immunohistochemistry (IHC) and/or fluorescent in situ hybridization (FISH) analysis of biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age;
2. Diagnosis of primary breast cancer with possible lymph node metastases before system (chemo+targeted therapy);
3. Availability of results from HER2 status previously determined on material from the primary tumor: HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive;
4. Sequential injection of 99mTc-ADAPT6 and 99mTc-DARPinG3 in the interval of 3-4 days in each HER2-positive breast cancer patient;
5. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
6. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination;
7. Subject is capable to undergo the diagnostic investigations to be performed in the study;
8. Informed consent

Exclusion Criteria:

1. Second, non-breast malignancy 2. Active current autoimmune disease or history of autoimmune disease 3. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C 5. Administration of other investigational medicinal product within 30 days of screening 6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with primary HER2-positive breast cancer
Enrollment: 15 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
99mTc-ADAPT6 uptake (counts)/SUV | 2 hours
  SPECT/CT-based 99mTc-ADAPT6 uptake value in primary tumor lesions (counts)/SUV of 99mTc-ADAPT6 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 2 hours after injection and measured in counts and SUV.
99mTc-ADAPT6 tumor-to-background ratio (SPECT) | 2 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-ADAPT6 uptake coinciding with tumor lesions (counts/SUV) will be divided by the value of 99mTc-ADAPT6 uptake coinciding with the regions without pathological findings (counts)
99mTc-DARPinG3 uptake (counts)/SUV | 4 hours
  SPECT/CT-based 99mTc-DARPinG3 uptake value in primary tumor lesions (counts)/SUV of 99mTc-DARPinG3 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 4 hours after injection and measured in counts and SUV
99mTc-DARPinG3 tumor-to-background ratio (SPECT) | 4 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-DARPinG3 uptake coinciding with tumor lesions (counts) will be divided by the value of 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (counts/the value of 99mTc-ADAPT6 and 99mTc-DARPinG3 uptake coinciding with tumor lesions (counts) will be divided by the value of 99mTc-ADAPT6 and 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (counts/SUV)
99mTc-ADAPT6 vs 99mTc-DARPinG3 uptake (counts)/SUV | 2 and 4 hours
  Comparison of SPECT/CT-based 99mTc-ADAPT6 versus 99mTc-DARPinG3 uptake value in primary tumor lesions (counts)/SUV of 99mTc-ADAPT6 and 99mTc-DARPinG3 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 2 and 4 hours after injection and measured in counts and SUV.
99mTc-ADAPT6 vs 99mTc-DARPinG3 tumor-to-background ratio (SPECT) | 2 and 4 hours
  Comparison of the value of 99mTc-ADAPT6 versus 99mTc-DARPinG3 uptake coinciding with tumor lesions (counts/SUV) divided by the value of 99mTc-ADAPT6 and 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (counts/SUV)

SECONDARY OUTCOMES:
99mTc-ADAPT6 vs immunohistochemical studies (percent) | 2 hours
  Sensitivity (%) of the method is assessed by comparing the 99mTc-ADAPT6 accumulation in the primary tumor with the results of immunohistochemical studies
99mTc-DARPinG3 vs immunohistochemical studies (percent) | 4 hours
  Sensitivity (%) of the method is assessed by comparing the 99mTc-DARPinG3 accumulation in the primary tumor with the results of immunohistochemical studies

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bragina, MD, Dsc, Principal Investigator — Tomsk NRMC
Locations (1):
- Tomsk NRMC, Tomsk, Russia